CLINICAL TRIAL: NCT03193099
Title: Decoding Presymptomatic White Matter Changes in Huntington Disease
Acronym: Win-HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C16-115; 2017-A00589-44 (Registry Identifier: RCB)
Record Dates: First submitted 2017-06-13; First posted 2017-06-20 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Huntington Disease; White Matter Alterations
MeSH Terms: conditions — Huntington Disease; Leukoaraiosis | interventions — Neuroimaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Premanifest HTT mutation carriers (Other)
  Interventions: Other: Brain imaging; Other: Neurological assessments; Behavioral: Psychological assessments; Behavioral: Behavioural assessments
- non HTT mutation carriers (Other)
  Interventions: Other: Brain imaging; Other: Neurological assessments; Behavioral: Psychological assessments; Behavioral: Behavioural assessments

INTERVENTIONS:
Other: Brain imaging — Volume, DWS and DTI
Other: Neurological assessments — UHDRS
Behavioral: Psychological assessments — STAI (Spielberger state and Trait Anxiety Inventory) A and B, BDI-II (Beck Depression Inventory), MINI (Mini-International Neuropsychiatric Interview) and MINI-SEA (mini Social cognitive and Emotional Assessment)
Behavioral: Behavioural assessments — Computerized game

SUMMARY:
WIN-HD is a monocentric longitudinal study comparing premanifest Huntingtin (HTT) mutation carriers and non HTT mutation carriers to determine that white-matter atrophy occurs far earlier than clinical onset in HD using Diffusion-weighted Nuclear Magnetic Resonance (N spectroscopy (DWS) and Diffusion Tensor Imaging (DTI).

The investigators will recruit up to 20 premanifest HTT mutation carriers (15 completed) and up to 20 non HTT mutation carriers (15 completed). It is important to have those 2 populations in order to compare our results and determine if there are significant white-matter changes far from the onset of HD. Therefore, non HTT mutation carriers will be age and gender matched to premanifest HTT mutation carriers.

In order to test the hypothesis, the study has 2 visits with a year interval.

This study is based on 4 principal criteria:

1. Imaging criteria
2. Clinical and neurological criteria
3. Psychological criteria
4. Behavioral criteria

ELIGIBILITY:
Inclusion Criteria:

* For presymptomatic individuals:

  * Genetic test available with CAG (Cytosine-Adenine-Guanine) repeat length > 36 in HTT gene
  * UHDRS score <5
  * Burden score <250
* For controls:

  - Genetic test available with CAG repeat length ≤ 36 in HTT gene
* Common inclusion criteria for presymptomatic individuals and controls (age-matched and gender-matched with presymptomatic individuals and but without any familial relationship):

  * At least 18 years of age
  * Capacity to consent
  * Signature of the informed consent
  * Covered by social security
  * Ability to undergo MRI scanning

Non-Inclusion Criteria:

* Under the age of 18 years of age
* Contra-indications to MRI examination (metallic implant, pacemaker, artificial heart valve, brain vascular malformation, aneurysm clips, exposed by metallic fragments, artificial implants, peripheral or neuronal stimulator, insulin pump, intravenous catheter, epilepsy, person with an history of seizure, metallic contraceptive device, permanent eyelid make up, claustrophobia,…)
* Unwillingness to be informed in case of abnormal MRI (with a significant medical anomaly)
* History of severe head injury
* History of neurological disorder or presence of neurological disorder
* Participation in a drug trial or exclusion period of another study
* Pregnancy or breastfeeding
* Inability to understand information about the protocol
* Person deprived of their liberty by judicial or administrative decision
* Person under legal protection (legal guardianship, tutelage or maintenance of justice)
* Person without any protection and unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Detection by Diffusion-weighted spectroscopy of abnormal white matter changes prior to the onset of Huntington disease comparing HTT mutation carriers and non HTT mutation carriers over one year | one year

SECONDARY OUTCOMES:
Detection by Diffusion-weighted spectroscopy of abnormal white matter changes over one year as an intersubject evolution | one year
Detection by Diffusion Tensor Imaging of abnormal white matter changes prior to the onset of Huntington disease comparing HTT mutation carriers and non HTT mutation carriers over one year. | one year
Detection by Diffusion Tensor Imaging white matter changes over one year as an intersubject evolution. | one year
Detection of abnormal scores from psychological tests to assess possible early non motor changes and their intersubject evolution over one year. | one year
Detection of choice rates and time differences in the behavioral task comparing HTT mutation carriers and non HTT mutation carriers over one year. | one year
Detection of time differences in the behavioral task comparing HTT mutation carriers and non HTT mutation carriers over one year. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra DURR, PU-PH, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Brain and Spine Institute, Paris, France

IPD SHARING:
Plan to Share IPD: No